CLINICAL TRIAL: NCT07356960
Title: Retrospective, Observational, Study on the Evaluation of the Real-world Outcome of Philadelphia-positive Acute Lymphoblastic Leukaemia Patients Treated With Ponatinib as First-line Treatment Under the Italian Law 648/96 (PONA4ALL Ph+)
Brief Title: Evaluation of the Efficacy of Ponatinib in Ph+ ALL in the Real-world
Acronym: PONA4ALL Ph+
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ALL3125
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphobkastic Leukemia; Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Keywords: ponatinib; real-world; philadelphia-positive acute lymphoblastic leukemia; Ph+ ALL; adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with ponatinib in first line: Patients treated with ponatinib as first line, alone or in combination with other antileukaemic agents, under Law 648/96.

SUMMARY:
The goal of this retrospective observational study is to learn about the efficacy of ponatinib in Philadelphia-positive ALL (Ph+ ALL) patients in a real-world setting. The main goal of the study is to assess the rate of complete molecular response (CMR) induced by ponatinib in patients treated under the regulations of Law 648/96, outside clinical trials.

Patients who were treated with ponatinib as part of their regular medical care and completed the follow-up period will be included in the study.

DETAILED DESCRIPTION:
This is a non-interventional, multicenter, strictly retrospective study including Ph+ ALL patients treated with ponatinib, alone or in combination with other antileukaemic agents, under Law 648/96. According to AIFA guideline 425-2024, all patients who received ponatinib as first-line treatment under Law 648/96 are eligible for inclusion provided that, at the time of enrolment, they are alive and have at least 18 months of retrospective observation available from the start of ponatinib treatment, or have died/lost to follow-up at any time after treatment initiation, regardless of the length of available follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years old;
2. Patient was treated in first-line with ponatinib monotherapy or in association with chemotherapy or immunotherapy;
3. Patient received ponatinib under the regulations of Law 648/96;
4. - Patient is alive and have at least 18 months of retrospective observation available from the start of ponatinib treatment, OR

   - has died/lost to follow-up at any time after treatment initiation, regardless of the length of available follow-up;
5. Signed informed consent, if applicable.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ph+ ALL patients treated with ponatinib, alone or in combination with other antileukaemic agents, under Law 648/96. According to AIFA guideline 425-2024, all patients who received ponatinib as first-line treatment under Law 648/96 are eligible for inclusion provided that, at the time of enrolment, they are alive and have at least 18 months of retrospective observation available from the start of ponatinib treatment, OR have died/lost to follow-up at any time after treatment initiation, regardless of the length of available follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2026-04-02 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ponatinib in terms of complete molecular response (CMR) achievement | 3 months
  Rate of patients treated with ponatinb in first-line who achieve complete molecular response (CMR) after induction

IPD SHARING:
Plan to Share IPD: No